CLINICAL TRIAL: NCT01497860
Title: Phase 2 Study of Weekly Vinorelbine in Children With Progressive or Recurrent Low-Grade Gliomas
Brief Title: Vinorelbine for Children With Progressive or Recurrent Low-grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eugene Hwang (Other)
Responsible Party: Sponsor-Investigator, Eugene Hwang, Assistant Professor, Pediatric Oncology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC-VRL
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-04

CONDITIONS: Low-grade Glioma
Keywords: pediatric; children; glioma; low-grade; vinorelbine; recurrent; progressive
MeSH Terms: conditions — Glioma; Recurrence | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine (Experimental): IV Vinorelbine (6mg/m2) provided once a week for 6 weeks followed by a 2 week rest (6 of every 8 weeks) for one year. Progression free survival will be monitored for 60 months.
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — IV Vinorelbine (6mg/m2) provided once a week for 6 weeks followed by a 2 week rest (6 of every 8 weeks) for one year. Progression free survival will be monitored for 60 months.
  Other Names: Navelbine

SUMMARY:
The purpose of this study is to investigate whether weekly Vinorelbine treatment can shrink or slow the growth of pediatric low-grade gliomas that have either returned or are continuing to grow.

Vinorelbine is a semi-synthetic vinca alkaloid that has recently generated interest in patients with pediatric low-grade glioma. It has been specifically synthesized to broaden its therapeutic spectrum and decrease the neurotoxicity associated with related agents.

DETAILED DESCRIPTION:
Different treatments exist for children with progressive or recurrent low-grade glioma. Each has variable efficacy at slowing or reversing growth, and exploration continues into finding better-tolerated, more effective treatments.

Vinorelbine has recently generated interest in stabilizing some pediatric low-grade gliomas. It has been fairly well tolerated in both adult and pediatric studies that have examined its use in other tumors.

Objective: To test the efficacy of Vinorelbine in children with pediatric low-grade glioma that has returned or continues to grow.

In this trial, Vinorelbine will be given intravenously once a week for 6 weeks followed by a 2 week rest (6 of every 8 weeks) for one year. The patients will then be followed for 60 months. Progression free survival is the primary outcome and defined as the none of the following: greater a 20% increase in the sun of the longest diameter of the target lesion, or a measurable increase in a non-target lesion, or the appearance of new lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age: < 18 years
* Tumor: Progressive or recurrent low grade glioma, WHO grade 1 or 2 who have failed at least one form of 'conventional' non-surgical therapy
* Histologic confirmation is required with the exception of optic pathway and brain stem gliomas. Patients are not required to have a re-operation at time of recurrence.
* Patients with disseminated disease are eligible.
* Children with neuro-fibromatosis and optic pathway or brainstem tumors are eligible but must have definitive radiologic or clinical evidence of progression
* Patients must have evidence of measureable disease
* Performance status: Karnofsky or Lansky performance status of >50%
* Organ Function:
* Adequate bone marrow function (ANC>1000/mm3, platelet count of >75,000/mm3, and hemoglobin > 8gm/dL) prior to starting therapy. Hemoglobin may be supported by transfusion
* Adequate liver function (SGPT/ALT<2.5 times ULN and bilirubin < 1.5 times ULN) prior to starting therapy
* Prior therapy:
* May have had treatment including surgery, chemotherapy, or radiotherapy for any number of relapses prior to enrollment
* Patients must have received their last fraction of radiotherapy >12 weeks prior to starting therapy
* Previous Vincristine or Vinblastine exposure is allowable.

Exclusion Criteria:

* No other significant medical illness that in the investigators' opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Any other cancer (except non-melanoma skin cancer), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* Patients of childbearing potential must not be pregnant or breast-feeding (vinorelbine is a pregnancy category D, no data on excretion in breastmilk)
* Patients of childbearing or fathering potential must practice adequate contraception

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2011-07; Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Hwang, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinorelbine: Patients with recurrent/progressive low-grade glioma, treatment six out of every eight weeks with IV vinorelbine for 12 months.
Period: Overall Study
Arm/Group | Vinorelbine
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vinorelbine: Patients with recurrent/progressive low-grade glioma, treatment six out of every eight weeks with IV vinorelbine for 12 months. Patients recruited without incidence over a 2 year period.
Arm/Group | Vinorelbine
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 6.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: IV Vinorelbine (6mg/m2) provided once a week for 6 weeks followed by a 2 week rest (6 of every 8 weeks) for one year. Progression free survival will be monitored for 60 months.
Time Frame: Assessed throughout the study from the first dose of the study drug to the date of progressive disease, death, or 60m.
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Vinorelbine
Number analyzed (Participants) | 13
percentage | 23.1 [14.8 to 31.1]

ADVERSE EVENTS:
Groups:
- Adverse Events: Neutropenia - Grade 4 (n=2) Thrombocytopenia - Grade 4 (n=1) Anemia - Grade 3 (n=2) Weight Loss - grade 2 (n=1)
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=13)
weight loss (General disorders) | 1 (1) — weight loss >10%
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 2 (3)
anemia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No